CLINICAL TRIAL: NCT00736658
Title: A Phase I, Randomised, Double-blind, Placebo-controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD1386 in Healthy Japanese Young and Elderly Subjects After Oral Multiple Doses.
Brief Title: AZD1386 Japanese Multiple Ascending Dosing Study
Acronym: JMAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Rolf Karlsten, MD, PhD, Medical Science Director Emerging Analgesia Clinical Neuroscience, AstraZeneca R&D Södertälje
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5090C00012
Record Dates: First submitted 2008-08-15; First posted 2008-08-18 (Estimated); Last update posted 2009-09-30 (Estimated); Status verified 2009-09

CONDITIONS: Chronic Pain
Keywords: Japanese; MAD; Multiple ascending dose; Chronic pain
MeSH Terms: conditions — Chronic Pain | interventions — AZD1386

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD1386 (Experimental): 4 groups receiving a specified volume of the active component AZD1386 at different points of time.
  Interventions: Drug: AZD1386
- Placebo (Placebo Comparator): Included in each dose group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1386 — Oral admin. of doses at 11 days through a 12 days period.
  Arms: AZD1386
Drug: Placebo — Oral admin. of doses at 11 days through a 12 days period.
  Arms: Placebo

SUMMARY:
This is a single centre, double-blind, randomised, parallel group, placebo controlled study to assess the safety, tolerability and pharmacokinetics of AZD1386 when given as multiple doses to 32 (24 healthy young and 8 healthy elderly) Japanese subjects. For young healthy subjects (aged ≥20 to ≤45 inclusive) 3 consecutive multiple ascending dose panels are planned. For elderly healthy subjects (aged ≥65 to≤80 inclusive) 1 multiple dose panel is planned.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese males or females young (≥20 to ≤45 years inclusive) or elderly (≥65 to ≤80 years inclusive). Female subjects must be surgically sterile or post-menopausal.
* Body Mass Index (BMI) of ≥19 to ≤ 27 kg/m2 and weight of ≥45 to ≤90 kg
* Clinically normal physical findings including heart rate > 45 bpm and laboratory values and normal resting ECG

Exclusion Criteria:

* History of somatic or psychiatric disease/condition, which may interfere with the objectives of the study as judged by the investigator
* A family history of short or long QT syndrome (SQTS) or sudden cardiac death (SCD) amongst first degree relatives
* Subjects with orthostatic hypotension defined as a decrease of ≥ 25mmHg systolic blood pressure and/or a decrease of ≥15mmHg diastolic blood pressure within 5 minutes when going from a supine to standing position
* Clinically significant illness or clinically relevant trauma within 2 weeks prior to the administration of the investigational product as judged by the investigator

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2008-06; Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To investigate the safety and tolerability of AZD1386 after multiple dosing in young and elderly healthy Japanese subjects by assessment of adverse events, vital signs, ECG parameters, body temperature, clinical chemistry, haematology and urinalysis. | All assessments are made at each visit during the study.

SECONDARY OUTCOMES:
To determine the PK profile of AZD1386 after multiple dosing by assessment of plasma concentrations. | Blood samples will be taken before and after study drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Karlsten, Study Director — Emerging Analgesia TA AstraZeneca R&D Södertälje, Sweden; Shunji Matsuki, Principal Investigator — Kyusyu Clinical Phramacology Research Clinic
Locations (1):
- Research Site, Fukuoka, Japan